CLINICAL TRIAL: NCT00164853
Title: Combined Sphincterotomy and Balloon Dilation (ESBD) Versus Standard Sphincterotomy (ES) in Removing Biliary Stones-a Randomized Controlled Trial
Brief Title: Compare Combined Sphincterotomy and Balloon Dilation (ESBD) Versus Standard Sphincterotomy (ES) in Removing Biliary Stones
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Anthony Yuen Bun Teoh, Department of Surgery, Chinese University of Hong Kong, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRE-2005.067-T
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2010-09

CONDITIONS: Common Bile Duct Stone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard sphincterotomy (ES) (Active Comparator): After deep cannulation, a pull-type sphincterotomy will be performed with a 25mm sphincterotome (eg clever cut, Olympus, Tokyo, Japan) with division of sphincter up to the duodenal wall. A complete sphincterotomy is defined by the free passage of a fully bowed sphincterotome with a 25m wire and spontaneous bile drainage.
  Interventions: Procedure: Standard sphincterotomy
- Sphincterotomy plus balloon dilation (ESBD) (Active Comparator): After complete sphincterotomy, a 3-cm long 15mm diameter CRE balloon is passed over a guidewire across the lower end of common bile duct. The contrast filled balloon is inflated to the size of the bile duct for around 30 seconds until waisting is abolished.
  Interventions: Procedure: endoscopic balloon dilatation

INTERVENTIONS:
Procedure: endoscopic balloon dilatation — Refer to description under arms
  Arms: Sphincterotomy plus balloon dilation (ESBD)
Procedure: Standard sphincterotomy — Refer to under arms
  Arms: Standard sphincterotomy (ES)

SUMMARY:
To compare the technique of combined balloon sphincter dilation after an initial sphincterotomy and standard sphincterotomy in the endoscopic removal of large bile duct stones. The investigators hypothesize that combined balloon dilation and sphincterotomy allows for easier stone removal without added morbidities when compared to standard sphincterotomy.

DETAILED DESCRIPTION:
Endoscopic sphincterotomy is a standard technique to enlarge the bile duct opening before stone removal during endoscopic retrograde cholangiopancreatography. However, complete sphincter ablation by endoscopic sphincterotomy is not always possible. Also, due to the tapering end of the distal duct, standard sphincterotomy may not be adequate for removal of particularly large stones. In a retrospective series by Ersoz et al, the addition of balloon dilation after sphincterotomy achieves a high stone clearance rate (89-95%). The investigators postulate that the combination of endoscopic sphincterotomy followed by balloon dilation may allow easier stone retrieval with acceptable complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old, presented to Prince of Wales Hospital for endoscopic retrograde cholangiopancreatography (ERCP) for known or suspected bile duct stones are invited to participate.
* Informed consent will be obtained before the beginning of ERCP.
* Patients are randomized to EST or ESBD after confirming the presence of bile duct stones on the initial cholangiogram

Exclusion Criteria:

* septic shock, coagulopathy (international normalized ratio >1.3,
* partial thromboplastin time greater than twice that of control),
* platelet count <50,000x103/uL or
* ampullary tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
stone clearance rate at the index session | 24 hours
  The ability to achieve complete stone clearance on the first ERCP

SECONDARY OUTCOMES:
Number of ERCP's required to achieve stone clearance | 3 months
  The number of ERCP procedures required to achieve complete stone clearance in the bile duct
ERCP related complications | 30 days
  These include complications that were described in consensus published in 1991

CONTACTS AND LOCATIONS:
Overall Officials: Frances KY Cheung, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Teoh AYB, Cheung FKY, Hu B, Pan YM, Lai LH, Chiu PWY, Wong SKH, Chan FKL, Lau JYW. Randomized trial of endoscopic sphincterotomy with balloon dilation versus endoscopic sphincterotomy alone for removal of bile duct stones. Gastroenterology. 2013 Feb;144(2):341-345.e1. doi: 10.1053/j.gastro.2012.10.027. Epub 2012 Oct 17. PMID 23085096